CLINICAL TRIAL: NCT03927443
Title: A Multi-Center, Evaluator -Masked, Randomized, Parallel Group, Active Controlled, Comparative Study of SPARC's SDP-133 Once Daily Compared With Lumigan ® 0.01% (Bimatoprost Ophthalmic Solution) in Subjects With Open Angle Glaucoma or Ocular Hypertension
Brief Title: A Comparative Study of SPARC's SDP-133 Once Daily and Lumigan in Subjects With Open Angle Glaucoma or Ocular Hypertension
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: [Sponsors decision]
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLR_17_21
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test (Experimental)
  Interventions: Drug: SDP-133
- Reference (Active Comparator)
  Interventions: Drug: Lumigan

INTERVENTIONS:
Drug: SDP-133 — one drop
  Arms: Test
Drug: Lumigan — one drop
  Arms: Reference

SUMMARY:
To evaluate the efficacy of once daily dosing with SPARC's novel ophthalmic formulation of bimatoprost compared with Lumigan 0.01% in subjects with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female, of 18 years of age or older
2. Provide signed and dated informed consent in accordance with good clinical practice (GCP) and local legislation prior to any study procedure.
3. Have open-angle glaucoma, (with or without pseudo exfoliation, pigment dispersion component) or ocular hypertension in both eyes and likely to be controlled on monotherapy.
4. Females of childbearing potential must not be pregnant or lactating (as confirmed by a negative urine pregnancy test Women of childbearing potential must agree to the use of a reliable method of contraception (e.g., total abstinence, intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], oral, transdermal, injected or implanted non- or hormonal contraceptive), throughout the study. A sterile sexual partner is not considered an adequate form of birth control. Subjects on hormonal contraceptives must have been on the same hormonal contraceptive for at least one month before the Screening and continue throughout the duration of the study. A female is considered of childbearing potential if she has had her first menses and she is either

   1. not postmenopausal for at least 12 consecutive months prior to enrollment;(Visit 1) or
   2. not surgically sterilized by bilateral tubal ligation, or bilateral oophorectomy, or hysterectomy
5. Male subjects with partners of childbearing potential who are not using birth control as described above must use a barrier method of contraception (eg. Condom) if not surgically sterile (ie, vasectomy).
6. Be able and willing to follow study instructions and complete all required visits.

Exclusion Criteria:

1. In the opinion of the investigator have uncontrolled or unstable systemic disease (eg, diabetes) which might interfere with the study. Subjects with a history of cancer or requiring cancer treatment within the past 5 years. Basal Cell and its treatment are allowed.
2. Current or history of subjects with depression, cerebral or active coronary insufficiency or orthostatic hypotension.
3. (If female of childbearing potential) Be pregnant, nursing, or planning a pregnancy from study entry and through the duration of the study.
4. In the opinion of the investigator the subject has clinically relevant, abnormally low or high blood pressure or pulse rate.
5. Have any known allergy or sensitivity to the study medications or their components.
6. Have any contraindications to bimatoprost therapy.
7. Be enrolled in an investigational drug or device study or have participated in such a study within 30 days prior to Visit 1.
8. Subject who may be involved in any aspect of the trial conduct, may not be an investigator, sub-investigator, or other site staff , or related to any site staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Mean Intra-ocular pressure (study eye) | Week 12.

SECONDARY OUTCOMES:
Time-matched change from baseline mean Intra-ocular pressure (study eye) | Week 12
Time-matched percent change in Intra-ocular pressure (study eye) | Week 12

OTHER OUTCOMES:
Adverse events | Week 13

IPD SHARING:
Plan to Share IPD: No